CLINICAL TRIAL: NCT04244331
Title: DETERMINATION OF THE CELL OF ORIGIN (COO) IN PATIENTS DIAGNOSED WITH DIFFUSE LARGE CELL B LYMPHOMA (LDCGB) IN SPANISH HOSPITALS OF GELTAMO GROUP
Brief Title: DETERMINATION OF THE CELL OF ORIGIN (COO) in LDCGB
Acronym: GELTAMO-COO
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Sponsor
Other Study IDs: GELTAMO-COO-2017-01
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2021-01

CONDITIONS: CCO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — TUMMORAL BIOPSIA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CCO — Determination of COO in tumor biopsies from patients with GBDD using the Lymph2Cx assay using NanoString tectology

SUMMARY:
This is a prospective, multicenter study, without any therapeutic intervention that will consist of the analysis of the results of the determination of the COO of all the patients diagnosed with LDCGB in the Spanish hospitals of GELTAMO that adhere to the project. The determination of the COO will be carried out prospectively at the Genomic Unit of the Hospital Clínic de Barcelona (IDIBAPS), where the histological samples of the patients will be sent for this purpose.

The main study variable will be the description of the COO (germ-center origin [GCB], activated [ABC], NOT DETERMINABLE, NOT VALUABLE)

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (LDCGB) is the most frequent form of lymphoma in Western countries, accounting for between 30 and 50% of all of them, and represents the paradigm of aggressive lymphoma (1). The current treatment is based on immunochemotherapy, that is, the combination of polychemotherapy (most commonly the CHOP regimen) with an anti-CD20 monoclonal antibody (rituximab). With this therapeutic approach a high proportion of patients are cured, but still 25-35% of them either do not respond to treatment or eventually relapse into the disease (2). New therapies in the experimental phase include other monoclonal antibodies of different specificity and small molecules with a target action.

LDCGB is actually heterogeneous and includes at least two subtypes depending on the cell of origin (COO): those related to a germline center B cell (GCB) and those similar to a post-germline center or activated B cell (ABC). Such groups show important biological, but also clinical and prognostic differences (3). Thus, ABC-type LDCGBs are more aggressive and patients have a worse prognosis. Recent data indicate that COO is also of therapeutic importance: thus, ABC-type LDCGBs would be particularly sensitive to NFkB and certain kinase inhibitors (4). Thus, the determination of COO now basically academic, is going to be a conventional diagnostic procedure in the coming years.

The determination of COO was initially carried out by a gene expression profiling (GEP) technique with frozen material (3). This technique is not realistic in the field of clinical care. Different immunohistochemical algorithms to mimic PEG results in paraffin tissue face great doubts about their reliability and, in fact, cannot be considered conventional (5). More recently, a NanoString technique has been implemented to determine the COO in paraffin tissue with an excellent correlation with PEG results (6). This technique has been used in the context of clinical trials, but no information is available in the general population setting. Precisely the aim of the present project is to apply the NanoString technique to the determination of COO of patients with LDCGB diagnosed during 2018 and 2019 in the Spanish centers associated to the cooperative group GELTAMO.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with LDCGB in the Spanish GELTAMO sites, without previous treatment and who decide to join the program.
* Age over or equal to 18 years old.
* Having voluntarily given informed consent for the sending and processing of biological samples, as well as for the analysis and reporting of the LDCGB COO results

Exclusion Criteria:

* Absence of histological material available to review histology and determine COO
* Patients with LDCGB from any other low-grade lymphoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with LDCGB an Age over or equal to 18 years old.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Develop Patform | 2 years
  The objective of the study is to develop a platform for the determination of the COO at a national level by means of NanoString in patients diagnosed with LDCGB and to analyze the distribution of this COO.

SECONDARY OUTCOMES:
Integration CCO | 2 years
  To analyze the feasibility of integrating prospective COO determination into clinical care practice.
Determination CCO | 15 days
  To determine the distribution of the COO (GCB, ABC or indeterminate) in the cases included in the LDCGB platform of the Spanish sites.

CONTACTS AND LOCATIONS:
Locations (1):
- GELTAMO, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No